CLINICAL TRIAL: NCT01851226
Title: Effect of Different Length of Time for Trainees to Attempt Cannulation on Success Rate of Selective Cannulation During hands-on ERCP Training
Acronym: ERCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20130415-3
Record Dates: First submitted 2013-05-04; First posted 2013-05-10 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Disease as Reason for ERCP

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 5 minutes group (Experimental): The time limit of attempt selective cannulation by trainees is limited to 5 minutes. If the trainees failed to enter the targeted duct within 5 minutes, the senior endoscopist would take over the duodenoscope and continue the following procedure of cannulation.
  Interventions: Procedure: Hands-on ERCP training.
- 10 minutes group (Experimental): The time limit of attempt selective cannulation by trainees is limited to 10 minutes. If the trainees failed to enter the targeted duct within 10 minutes, the senior endoscopist would take over the duodenoscope and continue the following procedure of cannulation.
  Interventions: Procedure: Hands-on ERCP training.
- 15 minutes group (Experimental): The time limit of attempt selective cannulation by trainees is limited to 15 minutes. If the trainees failed to enter the targeted duct within 15 minutes, the senior endoscopist would take over the duodenoscope and continue the following procedure of cannulation.
  Interventions: Procedure: Hands-on ERCP training.

INTERVENTIONS:
Procedure: Hands-on ERCP training. — The standard cannulation technique was used with a sphincterotome preloaded with a guidewire, positioned in the ampullary orifice, and targeting the presumed entry of common bile duct (CBD) or pancreatic duct (PD). During the whole procedure of cannulation by trainees, the senior endoscopist would actively communicate with trainees through verbal and/or hands-on assistance to help them to make the performance more correctly. If the trainees failed to enter the targeted duct within the designated length of time, the senior endoscopist would take over the duodenoscope and continue the following procedure of cannulation. The whole procedure of cannulation was recorded by video. Rectal indomethacin and/or pancreatic stent was used in high-risky patients.

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is one of the most difficult techniques in the field of GI endoscopy. It is necessary for trainees to spend enough time and perform enough cases to grasp this technique. The methods of ERCP training include hands-on teaching, training on different kinds of simulators, training on ex-vivo or live anesthetized porcine stomach models, etc. Supervised hands-on teaching is the standard method for ERCP training.

Selective cannulation is considered the most difficult and challenging part of learning ERCP. There is not an optimal time for trainees to attempt cannulation during hands-on ERCP training. The time used for attempting cannulation by trainees was 5min or 10min in several centers. In ERCP center of the investigators hospital, 15min was used for trainees to attempt cannulation for about one year. The incidence of post-ERCP pancreatitis, the major complication related to cannulation, was 4.0%, which was comparable with previous studies.

The investigators hypothesized that a longer time (15min) for trainees to attempt cannulation would increase success rate of selective cannulation and help to improve skills more quickly. At the meantime, with actively verbal or hands-on assistance from the instructor during performance of trainees, the risk of complications would not increased with a longer time to attempt cannulation. Here a prospective, endoscopists-blinded, randomized, controlled study was designed to evaluate the effects of different periods of time for trainees to attempt selective cannulation on success rate of cannulation, self-satisfaction of performance and post-ERCP pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 years old;
* Without prior EST.

Exclusion Criteria:

* History of partial or total gastrectomy (Billroth I/II, Roux-en-Y);
* Duodenal stricture (benign or malignant);
* Ampullary carcinoma;
* Previously failed selective cannulation;
* Chronic pancreatitis with PD stone;
* Minor papilla cannulation;
* Papilla fistula;
* Severe diseases of heart, lung, brain and kidney;
* Hemodynamical unstability;
* Pregnant women;
* Refusal or unable to give written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Success rate of selective cannulation by trainee | up to one year
  The rate of successful selective cannulation by trainee in one year.

SECONDARY OUTCOMES:
Complication rate | up to one year
  Post-ERCP pancreatitis (mild, moderate-to-severe); Abdominal pain (mild, moderate, severe); Hyperamylasemia; Vomiting (mild, moderate, severe); Cholangitis (mild, moderate, severe); Perforation (conservative therapy, surgery）; Bleeding (mild, moderate, severe);
Performance score of selective cannulation by trainees | up to one year
  How much will you score on your performance of cannulation? ----for trainee: 0-terrible, 10-perfect; How much will you score on the performance of cannulation by trainee? --for instructor: 0-terrible, 10-perfect.
Difficulty score of cannulation | up to one year
  How much will you score on the difficulty of the cannulation? -----for trainee: 0-very easy, 10-very difficult; How much will you score on the difficulty of the cannulation? -----for instructor: 0-very easy, 10-very difficult.
Final success rate of cannulation | up to one year
Total time of successful cannulation | up to one year
Rate of Needle-knife precut sphincterotomy | up to one year

CONTACTS AND LOCATIONS:
Overall Officials: Yanglin Pan, M.D., Principal Investigator — Associated professor
Locations (1):
- Endoscopic center, Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Swan MP, Alexander S, Moss A, Williams SJ, Ruppin D, Hope R, Bourke MJ. Needle knife sphincterotomy does not increase the risk of pancreatitis in patients with difficult biliary cannulation. Clin Gastroenterol Hepatol. 2013 Apr;11(4):430-436.e1. doi: 10.1016/j.cgh.2012.12.017. Epub 2013 Jan 11. PMID 23313840
- [Background] Nambu T, Ukita T, Shigoka H, Omuta S, Maetani I. Wire-guided selective cannulation of the bile duct with a sphincterotome: a prospective randomized comparative study with the standard method. Scand J Gastroenterol. 2011 Jan;46(1):109-15. doi: 10.3109/00365521.2010.521889. Epub 2010 Oct 6. PMID 20923377
- [Background] Tringali A, Mutignani M, Milano A, Perri V, Costamagna G. No difference between supine and prone position for ERCP in conscious sedated patients: a prospective randomized study. Endoscopy. 2008 Feb;40(2):93-7. doi: 10.1055/s-2007-995317. Epub 2007 Dec 5. PMID 18058651
- [Background] Testoni PA, Mariani A, Giussani A, Vailati C, Masci E, Macarri G, Ghezzo L, Familiari L, Giardullo N, Mutignani M, Lombardi G, Talamini G, Spadaccini A, Briglia R, Piazzi L; SEIFRED Group. Risk factors for post-ERCP pancreatitis in high- and low-volume centers and among expert and non-expert operators: a prospective multicenter study. Am J Gastroenterol. 2010 Aug;105(8):1753-61. doi: 10.1038/ajg.2010.136. Epub 2010 Apr 6. PMID 20372116
- [Background] Sutton VR, Hong MK, Thomas PR. Using the 4-hour Post-ERCP amylase level to predict post-ERCP pancreatitis. JOP. 2011 Jul 8;12(4):372-6. PMID 21737899
- [Background] Mariani A, Giussani A, Di Leo M, Testoni S, Testoni PA. Guidewire biliary cannulation does not reduce post-ERCP pancreatitis compared with the contrast injection technique in low-risk and high-risk patients. Gastrointest Endosc. 2012 Feb;75(2):339-46. doi: 10.1016/j.gie.2011.09.002. Epub 2011 Nov 9. PMID 22075192
- [Background] Kobayashi G, Fujita N, Imaizumi K, Irisawa A, Suzuki M, Murakami A, Oana S, Makino N, Komatsuda T, Yoneyama K. Wire-guided biliary cannulation technique does not reduce the risk of post-ERCP pancreatitis: multicenter randomized controlled trial. Dig Endosc. 2013 May;25(3):295-302. doi: 10.1111/j.1443-1661.2012.01372.x. Epub 2012 Sep 19. PMID 23368891
- [Derived] Pan Y, Zhao L, Leung J, Zhang R, Luo H, Wang X, Liu Z, Wan B, Tao Q, Yao S, Hui N, Fan D, Wu K, Guo X. Appropriate time for selective biliary cannulation by trainees during ERCP--a randomized trial. Endoscopy. 2015 Aug;47(8):688-95. doi: 10.1055/s-0034-1391564. Epub 2015 Mar 6. PMID 25750038